CLINICAL TRIAL: NCT00586443
Title: A Phase I Study of Bevacizumab, Everolimus, and Panitumumab for Patients With Advanced Solid Tumors
Brief Title: BEP Study Phase I (Bevacizumab, Everolimus, Panitumumab)
Acronym: BEP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Herbert Hurwitz, MD (Other)
Collaborators: Novartis (Industry); Genentech, Inc. (Industry); Amgen (Industry)
Responsible Party: Sponsor-Investigator, Herbert Hurwitz, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: Pro00001082
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Solid Tumors
Keywords: solid tumors; avastin; Phase I; Phase 1; combination therapy; bevacizumab; RAD001; everolimus; pantitumumab
MeSH Terms: interventions — Bevacizumab; Everolimus; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Other): This is a Phase I safety study. There is only one arm.
  Interventions: Drug: bevacizumab, everolimus, panitumumab

INTERVENTIONS:
Drug: bevacizumab, everolimus, panitumumab — Cohort # subjects Bevacizumab Everolimus Panitumumab
  * 3 3-6 5 mg/kg IV Q2 weeks 5 mg PO QoD 3.6 mg/kg IV Q2 weeks
  * 2 3-6 5 mg/kg IV Q2 weeks 5 mg PO QoD 4.8 mg/kg IV Q2 weeks
  * 1 3-6 10 mg/kg IV Q2 weeks 5 mg PO QD 4.8 mg/kg IV Q2 weeks
    1. 3-6 10 mg/kg IV Q2 weeks 10 mg PO QD 4.8 mg/kg IV Q2 weeks
    2. 3-6 10 mg/kg IV Q2 weeks 10 mg PO QD 6 mg/kg IV Q2 weeks 3a 10 RPTD* RPTD* RPTD* 3b 10 RPTD** RPTD** RPTD**
       * Panitumumab and RAD001 started on Day 1, bevacizumab started on Day 15. **Bevacizumab and RAD001 started on Day 1, panitumumab started on Day 15.
  Other Names: avastin; RAD001

SUMMARY:
Targeting molecular pathways of tumor growth has become a major focus of anti-cancer treatments. This study aims to investigate the toxicity, pharmacokinetics, and preliminary efficacy of the triplet combination of bevacizumab, RAD001, and panitumumab in patients with refractory solid tumors.

This open-labeled, non-randomized phase I trial of bevacizumab, everolimus and panitumumab is designed to assess the safety, tolerability and efficacy of this combination in adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
EGFr inhibition has been shown to have down-regulatory effects on VEGF expression and angiogenesis. The combination of anti-VEGF and anti-EGFr targeting is clinically rational, and preliminarily has shown at least additive, if not synergistic effects [12, 13]. Further, preclinical data has shown that constitutive activation of the AKT pathway is a mechanism of resistance to EGFr inhibitors [14]. Therefore, inhibition of both EGFr and AKT pathways by panitumumab and RAD001 may create a synergistic antitumor effect. There is also rationale that RAD001 and anti-VEGF therapies may be synergistic. Preliminary results from a Phase I dose escalation study of bevacizumab in combination with RAD001 has reported a recommended Phase II dose of this combination, and has described a minor response in a colorectal cancer patient previously refractory to bevacizumab-based therapy, and over 10 months of stable disease in another colorectal cancer patient previous refractory to bevacizumab-based therapy [15].

Bevicizumab (Avatstin) is a humanized monoclonal antibody to VEGF. VEGF is known to play a pivotal role in tumor angiogenesis and is a significant mitogenic stimulus for arterial, venous and lymphatic endothelial cells. The addition of bevacizumab to chemotherapy has been shown to increase overall response rate, duration of response and survival for patients with metastatic colon cancer (4) and is beneficial in first line non-small cell lung cancer and metastatic breast cancer [1, 2], and second line metastatic colorectal cancer (7). VEGF signals through phosphoatidylinositol 3-kinase (PI3K) and Akt as well as through the extracellular regulated kinase (ERK 1/2), a mitogen activated protein kinase (MAPK). VEGF's multiple biologic actions may be mediated by different pathways. Erikkson demonstrated that VEGF induced hyperpermeability was highly dependent on activation of the AKT pathway, while the angiogenic effect was largely unaffected by blocking this pathway and likely depended on ERK activation [3].

RAD001 (Everolimus), an oral derivative of rapamycin, selectively inhibits mTOR (mammalian target of rapamycin), an intracellular protein kinase implicated in the control of cellular proliferation of activated T-lymphocytes or neoplastic cells. mTOR is considered to be a downstream component of the PI3K/AKT/TSC pathway, a signalling module known to be heavily deregulated in many human cancers[4, 5]. In this context, there is an increasing body of evidence suggesting that AKT regulates mTOR activity[5-7], and that the activation status of the PI3K/AKT pathway may be indicative of responsiveness to rapamycins such as RAD001. Specifically, loss of PTEN or constitutive/hyper-activation of AKT has been suggested to sensitize tumors to the effects of inhibition of mTOR[6-8]. Indeed, RAD001 preferentially inhibits the proliferation of tumor cells displaying high AKT activity and totally reverses AKT-driven prostate intraepithelial neoplasia in a mouse transgenic model[7]. Rapamycins also inhibit downstream signaling pathways of VEGF. The rapamycin-regulated PI3K and p70s6 pathways are known to be involved in mediating VEGF's effects on endothelial cells [9]. In animal models, rapamycins modestly decrease tumor VEGF expression, and significantly blunt typical angiogenic responses to VEGF. Everolimus has been shown to inhibit tumor growth and reduce number of blood vessels in a murine melanoma model, indicating that RAD001 has direct antiangiogenic effects [10].

Panitumumab (Vectibix) is a fully humanized monoclonal antibody directed against epidermal growth factor receptor (EGFr), which is a 170-kD transmembrane glycoprotein with a cytoplasmic protein kinase domain essential for tumor growth and division. The receptor binds multiple ligands including epidermal growth factor and transforming growth factor-alpha (TGF-alpha). The tyrosine kinase intracellular domain of the receptor is activated via binding of a ligand to EGFr, which in turn initiates a cascade of intracellular signals. These downstream signaling pathways again include the phosphorylation of mitogen-activated protein kinase (MAPK) through the ras/raf pathway. Inhibition of these signaling pathways can result in cell growth arrest and apoptosis, respectively[11].

1. Sandler, A.B., et al. Randomized phase II/III trial of paclitaxel (P) plus carboplatin (C) with or without bevacizumab (NSC #704865) in patients with advanced non-squamous non-small cell lung cancer (NSCLC): An Eastern Cooperative Oncology Group (ECOG) Trial- E4599. in Proc Am Soc Clin Oncol. 2005.
2. Miller, K.D., et al. E2100: A randomized phase III trial of paclitaxel versus paclitaxel plus bevacizumab as first line threapy for locally recurrent or metastatic breast cancer. in American Society for Clinical Oncology. 2005. Orlando, FL.
3. Eriksson, A., et al., Small GTP-binding protein Rac is an essential mediator of vascular endothelial growth factor-induced endothelial fenestrations and vascular permeability. Circulation, 2003. 107(11): p. 1532-8.
4. Vivanco, I. and C.L. Sawyers, The phosphatidylinositol 3-kinase-akt pathway in human cancer. Nature Cancer, 2002. 2: p. 489-501.
5. Krymskaya, V.P., Tumor suppressors hamartin and tuberin: intracellular signaling. Cell Signal, 2003. 15: p. 729-739.
6. Bjornsti, M.-A. and P.J. Houghton, The TOR pathway: A target for cancer chemotherapy. Nat Rev Cancer, 2004. 4: p. 335-348.
7. Majumder, P.K., et al., mTOR inhibition reverses Akt-dependent prostate intraepithelial neoplasia through regulation of apoptotic and HIF-1-dependent pathways. Nat Med, 2004. 10: p. 594-601.
8. Noh, W.C., et al., Determinants of rapamycin in breast cancer cells. Clin Cancer Res, 2004. 10: p. 1013-1023.
9. Yu, Y. and J.D. Sato, MAP kinases, phosphatidylinositol 3-kinase, and p70 S6 kinase mediate the mitogenic response of human endothelial cells to vascular endothelial growth factor. J Cell Physiol, 1999. 178(2): p. 235-46.
10. Lane, H., et al. Antiangiogenic activity of RAD001, an orally active anticancer agent. in Proc AACR. 2002.
11. Ciardiello, F. and G. Tortora, A novel approach in the treatment of cancer: Targeting the epidermal growth factor receptor. Clin Cancer Res, 2001. 7: p. 2958-2970.
12. Spigel, D.R., et al. Bevacizumab and erlotinib in the treatment of patients with metastatic renal cell cancer (RCC): Update of a phase II multicenter trial. in Proc Am Soc Clin Oncol. 2005.
13. Saltz, L.B., et al. Randomized phase II trial of cetuximab/bevacizumab/irinotecan (CBI) versus cetuximab/bevacizumab (CB) in irinotecan-refractory colorectal cancer. in Proc Am Soc Clin Oncol. 2005.
14. She, Q.B., et al., Resistance to gefitinib in PTEN-null HER-overexpressing tumor cells can be overcome through restoration of PTEN function or pharmacologic modulation of constitutive phosphatidylinositol 3'-kinase/Akt pathway signaling. Clin Cancer Res, 2003. 9(12): p. 4340-6.
15. Zafar, Y., et al. Preliminary results of a phase I study of bevacizumab (BV) in combination with everolimus (E) in patients with advanced solid tumors. in Proc Am Soc Clin Oncol. 2006.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective. Disease must be measurable or evaluable by RECIST criteria.
* Patients must not have had radiation therapy, hormonal therapy, biologic therapy or chemotherapy for cancer within the 28 days prior to study day 1. Patients must not have had major surgery within the 28 days prior to study day 1 or minor surgical procedures within the 7 days prior to study day 1.
* Age >18 years.
* Karnofsky performance status > 70%.
* Life expectancy of at least 3 months.
* Patients must have normal organ and marrow function as defined below:

  **Absolute neutrophil count greater or equal to 1,500/μl; Platelets greater or equal to 100,000/μl; Total bilirubin, less or equal to 1.5 X upper limit of normal (ULN)AST(SGOT)/ALT(SGPT)less or equal to 2.5 X ULN less or equal to 5 X ULN if known hepatic metastases; Creatinine clearance greater or equal to 50 mL/min/m2 for patients with creatinine levels (by Cockroft-Gault equation or 24 hour urine; Hemoglobin > 9 g/dL; Magnesium > 1.2 mg/dL; Calcium (corrected for albumin)> 8.7 mg/dL
* The effect of the investigational drugs on the developing human fetus is not known, but these drugs are likely to be embryo- and feto- toxic. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study, she should inform her treating physician and study PI immediately. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had radiation therapy, hormonal therapy, biologic therapy, or chemotherapy for cancer within the 28 days prior to day 1 of the study.
* Patients who have received any other investigational agents within the 28 days prior to day 1 of the study.
* Patients with known CNS metastases or centrally-located non-small cell lung cancer.
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg)
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy. Patients on full dose anticoagulation are excluded from this trial.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment (56 days for hepatectomy, thoracotomy, neurosurgery) or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer, or bone fracture
* Proteinuria at screening as demonstrated by Urine protein:creatinine (UPC) ratio greater than 1.0
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* History of intolerance or hypersensitivity to prior treatment with bevacizumab, RAD001, or panitumumab. Prior treatment with these agents is otherwise permitted.
* Chronic treatment with systemic steroids or another immunosuppressive agent, though steroids may be used on an as-needed basis - ie - for treatment of nausea. Treatment with megace is permitted for treatment of anorexia.
* Other concurrent severe and/or uncontrolled medical disease which could compromise safety of treatment (i.e., severely impaired lung function, uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, ventricular arrhythmias, active ischemic heart disease, chronic liver or renal disease, active upper GI tract ulceration)
* A known history of HIV seropositivity, hepatitis C virus, acute or chronic active hepatitis B infection.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter drug absorption (e.g., inflammatory bowel disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or significant small bowel resection)
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumarin)
* Patients unwilling to or unable to comply with the protocol
* Medical need for the continued administration of any of the following drugs which affect CYP3A. (see Appendix A ifor a list of common medications).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit safety or compliance with study requirements or may interfere with the interpretation of the results.
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or any evidence of interstitial lung disease on baseline chest CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2007-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
To determine the MTD/recommended phase II regimen and evaluate safety of panitumumab added to RAD001 plus bevacizumab in adult patients with advanced solid tumors. | Every cycle (28-days)

SECONDARY OUTCOMES:
To preliminarily describe any clinical activity (PR, CR or duration of SD) associated with this regimen | Every cycle (28-days)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert I Hurwitz, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States